CLINICAL TRIAL: NCT04506203
Title: The Accuracy of Pediatric Air Test as a Non-invasive Atelectasis Diagnostic Tool: a Multi-centre Prospective Double-blind Study
Brief Title: The Accuracy of Pediatric Air Test as a Non-invasive Atelectasis Diagnostic Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Princesa (Unknown); Hospital Privado de Comunidad (Unknown)
Responsible Party: Principal Investigator, Patricio Gonzalez Pizarro, MD, PhD, Hospital Universitario La Paz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HULaPaz
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Lung Collapse; Lung Diseases; Atelectasis; Atelectasis Without Respiratory Distress Syndrome; Atelectases, Resorption; Air Test; Pediatric Disorder
Keywords: air test; atelectasis; pediatric; non-invasive; lung collapse
MeSH Terms: conditions — Pulmonary Atelectasis; Lung Diseases

STUDY DESIGN:
Masking Description: Lung Collapse will be diagnosed by a blind researcher that does not know the air test results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air test (Experimental)
  Interventions: Diagnostic Test: Air test

INTERVENTIONS:
Diagnostic Test: Air test — Patients will breathe 0.21 < FiO2 < 0.25 during 5 min and have a lung ultrasound perfomed at the end of the 5 min trial.

SUMMARY:
HYPOTHESIS:

During anesthetic pre-oxygenation with high FiO2, pulmonary atelectasis occur, especially in patients < 6 years old, where FRC and pulmonary closing volume may overlap. New borns and children <1 year old are especially vulnerable.

OBJECTIVES:

1. Validate "air test" as a individualized and non-invasive diagnostic method of clinically significant atelectasis in pediatrics.
2. Determine what other factors contribute to atelectasis development in pediatrics

METHODS:

30 pediatric patients will be studied with ages ranged between 45 postconceptional weeks and16 years old.

Baseline SpO2 and lung ultrasound will be performed for each patient upon arrival at the operating theatre before preoxygenation with FiO2 of 1.0 SpO2 will be measured 15 min after intubation during a 5 min long "air test" trial (FiO2 0.25). lung collapse will be verified by lung ultrasound at the end of the 15 min trial. Lung collapse will be eventually granted upon lung US verification by a blind researcher.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia
* Perioperative risk classification (ASA) I, II, III
* Newborns (postconceptional age> 45 weeks) to 16 years
* Need for oral / nasotracheal intubation

Exclusion Criteria:

* ASA > III
* Basal SpO2 < 97% on air in supine position
* Preoperative need for oxygen therapy and / or high-flow nasal cannulas
* Expected Difficult airway
* Presence of craniofacial disorders that may compromise ventilation
* Hemodynamic instability and / or need for inotropics
* History of untreated heart disease
* Presence or history of pneumothorax
* Presence of untreated congenital pulmonary disorders
* Refusal to participate in the study

Ages: 5 Weeks to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Atelectasis incidence | 5 minutes
  Assess incidence of SpO2 < 97% 15 minutes after anesthesia induction during a 5 minutes long air test (FiO2 < 0.25).
Accuracy of Pediatric Air test trial | 5 minutes
  Assess incidence of lung collapse (hence atelectasis incidence) 15 minutes after anesthesia induction using an air test (FiO2 < 0.25). Collapse blind validation using lung US

SECONDARY OUTCOMES:
Atelectasis risk factors assessment | 5 minutes
  Determine if there occurs higher atelectasis incidence depending on age, sex, medical records, body weight index or type of surgery
Atelectasis severity | 5 minutes
  Determine if there is any correlation between SpO2 values during air test and lung collapse, graded upon a validated severity lung collapse image score

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital Privado de Comunidad, Córdoba, Argentina
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD will be published in a peer reviewed journal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publishment in journal